CLINICAL TRIAL: NCT03615326
Title: A Phase III, Randomized, Double-blind Trial Comparing Trastuzumab Plus Chemotherapy and Pembrolizumab With Trastuzumab Plus Chemotherapy and Placebo as First-line Treatment in Participants With HER2 Positive Advanced Gastric or Gastroesophageal Junction Adenocarcinoma (KEYNOTE 811)
Brief Title: Pembrolizumab/Placebo Plus Trastuzumab Plus Chemotherapy in Human Epidermal Growth Factor Receptor 2 Positive (HER2+) Advanced Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma (MK-3475-811/KEYNOTE-811)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3475-811; MK-3475-811 (Other: MSD); 184142 (Registry Identifier: JAPAC-CTI); 2023-508253-98-00 (Registry Identifier: EU CT); U1111-1297-9360 (Registry Identifier: UTN); 2018-000224-34 (EudraCT Number)
Record Dates: First submitted 2018-07-31; First posted 2018-08-03 (Actual); Results first posted 2025-03-17 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Gastric Neoplasms; Gastroesophageal Junction Adenocarcinoma
Keywords: programmed cell death receptor 1 (PD-1); programmed cell death ligand 1 (PD-L1); anti-PD-1; anti PD-1; GEJ; Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Cisplatin; Fluorouracil; Oxaliplatin; Capecitabine; S 1 (combination); Trastuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Global Pembrolizumab + Standard of Care First Course (Experimental): Participants received 200 mg pembrolizumab IV every 3 weeks (Q3W) plus trastuzumab (8 mg/kg loading dose, 6 mg/kg maintenance thereafter) IV Q3W in combination with investigator's choice of FP or CAPOX chemotherapy.
  Interventions: Biological: Pembrolizumab; Drug: Cisplatin; Drug: 5-FU; Drug: Oxaliplatin; Drug: Capecitabine; Biological: Trastuzumab
- Global Standard of Care (Active Comparator): Participants received matched placebo to pembrolizumab IV Q3W plus trastuzumab (8mg/kg loading dose, 6mg/kg maintenance thereafter) IV Q3W in combination with investigator's choice of FP or CAPOX chemotherapy.
  Interventions: Biological: Placebo; Drug: Cisplatin; Drug: 5-FU; Drug: Oxaliplatin; Drug: Capecitabine; Biological: Trastuzumab
- Japan Pembrolizumab + Trastuzumab + S-1 Plus Oxaliplatin (Experimental): Participants received 200 mg pembrolizumab IV every 3 weeks (Q3W) plus trastuzumab (8 mg/kg loading dose, 6 mg/kg maintenance thereafter) IV Q3W in combination with SOX chemotherapy.
  Interventions: Biological: Pembrolizumab; Drug: Oxaliplatin; Drug: S-1; Biological: Trastuzumab
- Japan Trastuzumab + S-1 Plus Oxaliplatin (Experimental): Participants received matched placebo to pembrolizumab IV Q3W plus trastuzumab (8mg/kg loading dose, 6mg/kg maintenance thereafter) IV Q3W in combination with SOX chemotherapy.
  Interventions: Biological: Placebo; Drug: Oxaliplatin; Drug: S-1; Biological: Trastuzumab

INTERVENTIONS:
Biological: Pembrolizumab — 200 mg on Day 1 of each 3-week cycle as an IV infusion.
  Other Names: Keytruda®; MK-3475
  Arms: Global Pembrolizumab + Standard of Care First Course; Japan Pembrolizumab + Trastuzumab + S-1 Plus Oxaliplatin
Biological: Placebo — Solution for IV infusion on Day 1 of each 3-week cycle.
  Arms: Global Standard of Care; Japan Trastuzumab + S-1 Plus Oxaliplatin
Drug: Cisplatin — 80 mg/m^2 on Day 1 of each 3-week cycle as an IV infusion, administered as part of FP chemotherapy regimen.
  Arms: Global Pembrolizumab + Standard of Care First Course; Global Standard of Care
Drug: 5-FU — 800 mg/m^2/day continuous on Days 1-5 of each 3-week cycle (120 hours or per local standard), administered as part of FP chemotherapy regimen.
  Arms: Global Pembrolizumab + Standard of Care First Course; Global Standard of Care
Drug: Oxaliplatin — 130 mg/m^2 on Day 1 of each 3-week cycle over 2 hours as an IV infusion, administered as part of CAPOX chemotherapy regimen and as part of SOX chemotherapy regimen.
Drug: Capecitabine — 1000 mg/m^2 as oral capsules BID on Days 1-14 of each 3-week cycle, administered as part of CAPOX chemotherapy regimen.
  Arms: Global Pembrolizumab + Standard of Care First Course; Global Standard of Care
Drug: S-1 — Combination product of tegafur, CDHP, and Oxo. Oral capsules BID on Days 1-14 of each 3-week cycle based on body surface area (BSA): <1.25 m^2 BSA =40 mg, 1.25 to <1.5 m^2 BSA=50 mg, ≥1.5 m^2 BSA=60 mg. Administered as part of SOX chemotherapy regimen.
  Arms: Japan Pembrolizumab + Trastuzumab + S-1 Plus Oxaliplatin; Japan Trastuzumab + S-1 Plus Oxaliplatin
Biological: Trastuzumab — 8 mg/kg loading dose and then 6 mg/kg maintenance dose administered IV on day 1 of each 3-week cycle.
  Other Names: Herceptin®

SUMMARY:
The study will compare the efficacy and safety of pembrolizumab plus trastuzumab in combination with standard of care (SOC) chemotherapy versus trastuzumab in combination with SOC chemotherapy in participants with HER2-positive gastric cancer. The primary hypotheses of the study are that pembrolizumab plus trastuzumab in combination with chemotherapy is superior to trastuzumab plus chemotherapy in terms of 1) progression free survival (PFS) per Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) as assessed by blinded independent central review (BICR), and 2) overall survival (OS).

DETAILED DESCRIPTION:
Pembrolizumab (200 mg) or placebo will be administered intravenously [IV] on day 1 of each 3-week cycle. Trastuzumab (8 mg/kg loading dose, 6 mg/kg maintenance dose) will be administered IV on day 1 of each 3-week cycle. SOC chemotherapy for the global cohort will either be FP (80 mg/m^2 cisplatin administered IV on Day 1 of each 3-week cycle and 800 mg/m^2 5-fluorouracil [5-FU] administered IV on Days 1-5 of each 3-week cycle) or CAPOX (1000 mg/m^2 capecitabine administered orally twice daily [BID] on days 1-14 of each 3-week cycle and 130 mg/m^2 oxaliplatin administered IV on Day 1 of each 3-week cycle). A Japan cohort will receive SOX chemotherapy consisting of S-1 (tegafur, 5-chloro-2,4-dihydroxypyridine [CDHP], and potassium oxonate [Oxo]) administered orally BID according to Body Surface Area (BSA) on Days 1-14 of each 3-week cycle and oxaliplatin (130 mg/m^2) administered IV on Day 1 each 3-week cycle.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria include, but are not limited to:

* Histologically or cytologically confirmed diagnosis of previously untreated, locally advanced unresectable or metastatic human epidermal growth factor receptor 2 (HER2) positive gastric or gastroesophageal junction (GEJ) adenocarcinoma
* HER2-positive defined as either immunohistochemistry (IHC) 3+ or IHC 2+ in combination with in-situ hybridization positive (ISH+) or fluorescent in-situ hybridization (FISH), as assessed by central review on primary or metastatic tumor
* Has measurable disease as defined by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as determined by the site investigator
* Male participants must agree to use approved contraception
* Female participants who are not pregnant or breastfeeding, and who are either not a woman of childbearing potential (WOCBP), or are a WOCBP who agrees to use approved contraception
* Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale within 3 days prior to the first dose of trial treatment
* Has a life expectancy of greater than 6 months
* Has adequate organ function

Exclusion Criteria:

Exclusion criteria include, but are not limited to:

* Has had previous therapy for locally advanced unresectable or metastatic gastric/GEJ cancer
* Has had major surgery, open biopsy or significant traumatic injury within 28 days prior to randomization, or anticipation of the need for major surgery during the course of study treatment
* Has had radiotherapy within 14 days of randomization
* Has a known additional malignancy that is progressing or has required active treatment within the past 5 years
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Has a known history of active tuberculosis (TB; Mycobacterium tuberculosis)
* Has an active infection requiring systemic therapy
* Has poorly controlled diarrhea
* Accumulation of pleural, ascitic, or pericardial fluid requiring drainage or diuretic drugs within 2 weeks prior to enrollment. If the participant is receiving diuretic drugs for other reasons, it is acceptable
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the participant's participation for the full duration of the trial, or is not in the best interest of the participant to participate, in the opinion of the treating investigator
* Has peripheral neuropathy > Grade 1
* Has a known psychiatric or substance abuse disorder that would interfere with cooperation with the requirements of the trial
* A WOCBP who has a positive urine pregnancy test within 24 hours prior to randomization or treatment allocation
* Has active or clinically significant cardiac disease
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies)
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab, trastuzumab, study chemotherapy agents and/or to any excipients, murine proteins, or platinum-containing products
* Has had an allogeneic tissue/solid organ transplant
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], OX 40, Cluster of Differentiation 137 [CD137])

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 738 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2025-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (192):
- United States (23):
  - UCLA Hematology/Oncology - Westwood (Building 200 Suite 120) ( Site 0045), Los Angeles, California
  - Pacific Cancer Care ( Site 0063), Monterey, California
  - UC Irvine Medical Center/Chao Family Comprehensive Cancer Center ( Site 0050), Orange, California
  - University of Miami Sylvester Comprehensive Cancer Center - Plantation ( Site 0026), Miami, Florida
  - Southeastern Regional Medical Center, Inc. ( Site 0058), Newnan, Georgia
  - Midwestern Regional Medical Center, Inc. ( Site 0059), Zion, Illinois
  - Beth Israel Deaconess Medical Center ( Site 0070), Boston, Massachusetts
  - Dana-Farber Cancer Institute [Boston, MA] ( Site 0010), Boston, Massachusetts
  - Minnesota Oncology Hematology, PA ( Site 8001), Minneapolis, Minnesota
  - Washington University School of Medicine ( Site 0040), St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center- Monmouth ( Site 0071), Middletown, New Jersey
  - Memorial Sloan-Kettering Cancer Center at West Harrison ( Site 0065), Harrison, New York
  - Memorial Sloan-Kettering Cancer Center ( Site 0017), New York, New York
  - University of Rochester ( Site 0041), Rochester, New York
  - Levine Cancer Institute ( Site 0015), Charlotte, North Carolina
  - Duke Cancer Institute ( Site 0042), Durham, North Carolina
  - CTCA Southwestern ( Site 0060), Tulsa, Oklahoma
  - Cancer Treatment Centers of America-Eastern Regional Medical Center ( Site 0025), Philadelphia, Pennsylvania
  - Allegheny General Hospital ( Site 0053), Pittsburgh, Pennsylvania
  - Sanford Hematology Oncology-Sioux Falls SD ( Site 0004), Sioux Falls, South Dakota
  - University of Texas MD Anderson Cancer Center ( Site 0001), Houston, Texas
  - Oncology & Hematology Assoc. SW Virginia, Inc., DBA Blue Ridge Cancer Care ( Site 8000), Roanoke, Virginia
  - Seattle Cancer Care Alliance ( Site 0038), Seattle, Washington
- Australia (4):
  - Liverpool Hospital ( Site 2206), Liverpool, New South Wales
  - Westmead Hospital ( Site 2200), Westmead, New South Wales
  - Southern Medical Day Care Centre ( Site 2207), Wollongong, New South Wales
  - Monash Health ( Site 2202), Clayton, Victoria
- Brazil (8):
  - Instituto do Cancer do Ceara ( Site 0208), Fortaleza, Ceará
  - Hospital Sao Rafael ( Site 0209), Salvador, Estado de Bahia
  - CIONC - Centro Integrado de Oncologia de Curitiba ( Site 0205), Curitiba, Paraná
  - Hospital de Caridade de Ijui ( Site 0202), Ijuí, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao ( Site 0203), Porto Alegre, Rio Grande do Sul
  - CEPON - Centro de Pesquisas Oncologicas ( Site 0200), Florianópolis, Santa Catarina
  - Instituto Nacional do Cancer Jose Alencar Gomes da Silva INCA ( Site 0201), Rio de Janeiro
  - IBCC - Instituto Brasileiro de Controle do Cancer ( Site 0204), São Paulo
- Chile (5):
  - Clinica Universidad Catolica del Maule ( Site 0305), Talca, Maule Region
  - Fundacion Arturo Lopez Perez FALP ( Site 0302), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile ( Site 0301), Santiago, Region M. de Santiago
  - Instituto Nacional del Cancer ( Site 0303), Santiago, Region M. de Santiago
  - Centro Investigación del Cáncer James Lind ( Site 0300), Temuco, Región de la Araucanía
- China (19):
  - Shanghai General Hospital ( Site 2404), Shanghai, Anhui
  - Peking Union Medical College Hospital ( Site 2419), Beijing, Beijing Municipality
  - Fifth Medical Center of CPLA General Hospital ( Site 2415), Beijing, Beijing Municipality
  - Beijing Cancer Hospital ( Site 2413), Beijing, Beijing Municipality
  - Fujian Provincial Cancer Hospital ( Site 2418), Fuzhou, Fujian
  - 900 Hospital of the Joint ( Site 2420), Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University ( Site 2431), Xiamen, Fujian
  - Guangdong General Hospital ( Site 2433), Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital ( Site 2407), Harbin, Heilongjiang
  - Henan Cancer Hospital ( Site 2400), Zhengzhou, Henan
  - Xiangya Hospital Central-South University ( Site 2426), Changsha, Hunan
  - Jiangsu Cancer Hospital ( Site 2432), Nanjing, Jiangsu
  - The First Hospital Of Jilin University ( Site 2402), Changchun, Jilin
  - Fudan University Shanghai Cancer Center ( Site 2424), Shanghai, Shanghai Municipality
  - Zhongshan Hospital affiliated to Fudan University ( Site 2401), Shanghai, Shanghai Municipality
  - Cancer Hospital Affiliated to Xinjiang Medical University ( Site 2430), Ürümqi, Xinjiang
  - The First Affiliated Hospital.Zhejiang University ( Site 2408), Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital ( Site 2412), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital ( Site 2409), Hangzhou, Zhejiang
- France (9):
  - CHU de Rouen ( Site 0912), Rouen, Ain
  - HUS Hopital Hautepierre ( Site 0910), Strasbourg, Bas-Rhin
  - Hopital Jean Minjoz Besancon ( Site 0901), Besançon, Doubs
  - C.H.R.U. de Brest - Hopital Morvan ( Site 0913), Brest, Finistere
  - Centre Oscar Lambret ( Site 0911), Lille, Nord
  - Centre Leon Berard ( Site 0904), Lyon, Rhone
  - Institut de Cancerologie de l Ouest Centre Rene Gauducheau ( Site 0902), Saint-Herblain, Val-de-Marne
  - Institut Gustave Roussy ( Site 0900), Villejuif, Val-de-Marne
  - CHU Hopital Saint Antoine ( Site 0905), Paris
- Germany (11):
  - SLK-Kliniken Heilbronn ( Site 1015), Heilbronn, Baden-Wurttemberg
  - Klinikum Ludwigsburg ( Site 1014), Ludwigsburg, Baden-Wurttemberg
  - Innere Medizin I, Universitaetsklinikum Tuebingen ( Site 1020), Tübingen, Baden-Wurttemberg
  - Klinikum rechts der Isar der Technischen Universitaet ( Site 1027), Munich, Bavaria
  - Medizinische Hochschule Hannover ( Site 1019), Hanover, Lower Saxony
  - Universitaetsklinikum Carl Gustav Carus der Technischen Univ ( Site 1001), Dresden, Saxony
  - Universitaetsklinikum Leipzig AOeR ( Site 1007), Leipzig, Saxony
  - Charite-Universitaetsmedizin Berlin Campus Virchow-Klinikum ( Site 1026), Berlin
  - Klinikum Bremen Nord ( Site 1017), Bremen
  - Facharztzentrum Eppendorf ( Site 1025), Hamburg
  - Asklepios Klinik Altona ( Site 1000), Hamburg
- Guatemala (6):
  - Celan SA ( Site 0504), Guatemala City
  - Oncomedica ( Site 0500), Guatemala City
  - Grupo Angeles SA ( Site 0501), Guatemala City
  - Nucare Center ( Site 0506), Guatemala City
  - Medi-K Cayala ( Site 0505), Guatemala City
  - Centro Regional de Sub Especialidades Medicas SA ( Site 0502), Quetzaltenango
- Ireland (3):
  - Saint James's Hospital ( Site 1505), Dublin
  - Beaumont Hospital ( Site 1506), Dublin
  - Tallaght University Hospital ( Site 1513), Dublin
- Israel (8):
  - Soroka University Medical Center ( Site 1603), Beersheba
  - Rambam Health Care Campus ( Site 1606), Haifa
  - Edith Wolfson Medical Center ( Site 1605), Holon
  - Hadassah Ein Kerem Medical Center ( Site 1604), Jerusalem
  - Meir Medical Center ( Site 1609), Kfar Saba
  - Rabin Medical Center ( Site 1602), Petah Tikva
  - Chaim Sheba Medical Center. ( Site 1607), Ramat Gan
  - Sourasky Medical Center ( Site 1601), Tel Aviv
- Italy (8):
  - AUOP Ospedale Santa Chiara ( Site 1100), Pisa, Tuscany
  - Humanitas Gavazzeni ( Site 1106), Bergamo
  - Universita Magna Graecia di Catanzaro ( Site 1107), Catanzaro
  - IEO Istituto Europeo di Oncologia ( Site 1105), Milan
  - Azienda Ospedaliero - Universitaria Policlinico di Modena ( Site 1102), Modena
  - A.O.U. Universita degli Studi della Campania-Luigi Vanvitelli ( Site 1103), Napoli
  - Istituto Oncologico Veneto ( Site 1101), Padua
  - Ospedale Civile Spirito Santo ( Site 1104), Pescara
- Japan (30):
  - Aichi Cancer Center Hospital ( Site 2617), Nagoya, Aichi-ken
  - National Cancer Center Hospital East ( Site 2605), Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center ( Site 2615), Matsuyama, Ehime
  - Gunma Prefectural Cancer Center ( Site 2602), Ohta, Gunma
  - Hyogo Cancer Center ( Site 2619), Akashi, Hyōgo
  - Kobe City Medical Center General Hospital ( Site 2614), Kobe, Hyōgo
  - Ibaraki Prefectural Central Hospital ( Site 2611), Kasama, Ibaraki
  - Kagawa University Hospital ( Site 2604), Kita-gun, Kagawa-ken
  - Kanagawa Cancer Center ( Site 2603), Yokohama, Kanagawa
  - Osaki Citizen Hospital ( Site 2626), Ōsaki, Miyagi
  - Kansai Medical University Hospital ( Site 2618), Hirakata, Osaka
  - Kindai University Hospital ( Site 2616), Sayama, Osaka
  - Osaka University Hospital ( Site 2600), Suita, Osaka
  - Saitama Cancer Center ( Site 2620), Kitaadachi-gun, Saitama
  - Shizuoka Cancer Center Hospital and Research Institute ( Site 2607), Sunto-gun, Shizuoka
  - Tochigi Cancer Center ( Site 2627), Utsunomiya, Tochigi
  - Kyorin University Hospital ( Site 2608), Mitaka, Tokyo
  - Chiba Cancer Center ( Site 2623), Chiba
  - National Hospital Organization Kyushu Cancer Center ( Site 2609), Fukuoka
  - Gifu University Hospital ( Site 2621), Gifu
  - Hiroshima City Hiroshima Citizens Hospital ( Site 2625), Hiroshima
  - Kumamoto University Hospital ( Site 2601), Kumamoto
  - Niigata Cancer Center Hospital ( Site 2622), Niigata
  - National Hospital Organization - Osaka National Hospital - Institute For Clinical Research ( Site 26, Osaka
  - Osaka International Cancer Institute ( Site 2613), Osaka
  - Osaka General Medical Center ( Site 2624), Osaka
  - National Cancer Center Hospital ( Site 2612), Tokyo
  - Toranomon Hospital ( Site 2628), Tokyo
  - Tokyo Metropolitan Komagome Hospital ( Site 2606), Tokyo
  - The Cancer Institute Hospital of JFCR ( Site 2610), Tokyo
- Auckland City Hospital ( Site 2300), Auckland, New Zealand
- Poland (8):
  - Przychodnia Lekarska Komed ( Site 1716), Konin, Greater Poland Voivodeship
  - Uniwersytecki Szpital Kliniczny im. J. M. Radeckiego we Wroclawiu ( Site 1705), Wroclaw, Lower Silesian Voivodeship
  - Dolnoslaskie Centrum Onkologii. ( Site 1712), Wroclaw, Lower Silesian Voivodeship
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 w Lublinie ( Site 1709), Lublin, Lublin Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie (, Warsaw, Masovian Voivodeship
  - Szpital Morski im. PCK. Szpitale Pomorskie Sp. Z o.o ( Site 1715), Gdynia, Pomeranian Voivodeship
  - Szpital Specjalistyczny w Koscierzynie Sp. z o.o. ( Site 1708), Kościerzyna, Pomeranian Voivodeship
  - Beskidzkie Centrum Onkologii im. Jana Pawla II ( Site 1710), Bielsko-Biala, Silesian Voivodeship
- Russia (8):
  - Republican Clinical Oncology Dispensary of Republic of Bashkortostan ( Site 1807), Ufa, Baskortostan, Respublika
  - Chelyabinsk Regional Clinical Oncological Dispensary ( Site 1815), Chelyabinsk, Chelyabinsk Oblast
  - Blokhin National Medical Oncology ( Site 1805), Moscow, Moscow
  - Podolsky City Clinical Hospital ( Site 1817), Podolsk, Moscow Oblast
  - Medical University REAVIZ ( Site 1816), Samara, Samara Oblast
  - Leningrad Regional Oncology Center ( Site 1800), Saint Petersburg, Sankt-Peterburg
  - Scientific Research Oncology Institute n.a. N.N.Petrov ( Site 1801), Saint Petersburg, Sankt-Peterburg
  - St Petersburg City Clinical Oncology Dispensary ( Site 1812), Saint Petersburg, Sankt-Peterburg
- South Korea (4):
  - Seoul National University Hospital ( Site 2703), Seoul
  - Severance Hospital Yonsei University Health System ( Site 2700), Seoul
  - Asan Medical Center ( Site 2702), Seoul
  - Samsung Medical Center ( Site 2701), Seoul
- Spain (7):
  - Hospital General Universitario de Elche ( Site 1404), Elche, Alicante
  - Hospital Germans Trias i Pujol. ICO de Badalona ( Site 1410), Badalona, Barcelona
  - Hospital Universitario Marques de Valdecilla ( Site 1405), Santander, Cantabria
  - Hospital Universitario Quiron Madrid ( Site 1407), Pozuelo de Alarcón, Madrid
  - Hospital Universitario Central de Asturias ( Site 1402), Oviedo, Principality of Asturias
  - Hospital General Universitari Vall d Hebron ( Site 1401), Barcelona
  - Hospital Universitario Ramon y Cajal ( Site 1400), Madrid
- Turkey (Türkiye) (9):
  - Adana Sehir Hastanesi ( Site 2002), Adana
  - Hacettepe Universitesi Tip Fakultesi Hastanesi ( Site 2017), Ankara
  - Abdurrahman Yurtaslan Onkoloji Egitim ve Arastirma Hastanesi ( Site 2006), Ankara
  - Trakya Universitesi Tip Fakultesi ( Site 2015), Edirne
  - Ataturk Universitesi Tip Fakultesi Hastanesi ( Site 2000), Erzurum
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi ( Site 2001), Istanbul
  - Dokuz Eylul Universitesi Tip Fakultesi Hastanesi ( Site 2011), Izmir
  - Malatya Inonu Universitesi Tip Fakultesi Hastanesi ( Site 2009), Malatya
  - Sakarya Universitesi Egitim ve Arastirma Hastanesi ( Site 2012), Sakarya
- Ukraine (11):
  - City Clinical Hosp.4 of DCC ( Site 2102), Dnipro, Dnipropetrovsk Oblast
  - MI Kryviy Rih Center of Dnipropetrovsk Regional Council ( Site 2101), Kryviy Rih, Dnipropetrovsk Oblast
  - MI Precarpathian Clinical Oncology Center ( Site 2105), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Communal non profit enterprise Regional Clinical Oncology Center ( Site 2112), Kharkiv, Kharkivs’ka Oblast’
  - Medical Center Asklepion LLC ( Site 2115), Khodosovka, Kyivska Oblast
  - Clinic of National Cancer Institute ( Site 2104), Kyiv, Kyivska Oblast
  - Medical and Diagnostic Centre LLC Dobryi Prognoz ( Site 2114), Kyiv, Kyivska Oblast
  - Lviv State Oncology Regional Treatment and Diagnostic Center ( Site 2106), Lviv, Lviv Oblast
  - MI Odessa Regional Oncological Centre ( Site 2108), Odesa, Odesa Oblast
  - Medical Centre LLC Oncolife ( Site 2103), Zaporizhzhya, Zaporizhzhia Oblast
  - Kyiv City Clinical Oncology Centre ( Site 2110), Kyiv
- United Kingdom (10):
  - Royal Hospital in Derby ( Site 1514), Derby, Derbyshire
  - Ninewells Hospital and Medical School ( Site 1504), Dundee, Dundee City
  - Castle Hill Hospital ( Site 1501), Cottingham, East Riding Of Yorkshire
  - University College London Hospital NHS Foundation Trust ( Site 1508), London, London, City of
  - St Georges University Hospitals NHS Foundation Trust. ( Site 1500), London, London, City of
  - Royal Marsden Hospital ( Site 1510), Sutton, Surrey
  - Royal Marsden NHS Foundation Trust ( Site 1512), London
  - The Christie Hospital NHS Foundation Trust ( Site 1503), Manchester
  - Mount Vernon Cancer Centre ( Site 1507), Northwood
  - Manor Hospital Walsall England ( Site 1515), Walsall

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Janjigian YY, Kawazoe A, Bai Y, Xu J, Lonardi S, Metges JP, Yanez P, Wyrwicz LS, Shen L, Ostapenko Y, Bilici M, Chung HC, Shitara K, Qin SK, Van Cutsem E, Tabernero J, Li K, Shih CS, Bhagia P, Rha SY; KEYNOTE-811 Investigators. Pembrolizumab plus trastuzumab and chemotherapy for HER2-positive gastric or gastro-oesophageal junction adenocarcinoma: interim analyses from the phase 3 KEYNOTE-811 randomised placebo-controlled trial. Lancet. 2023 Dec 9;402(10418):2197-2208. doi: 10.1016/S0140-6736(23)02033-0. Epub 2023 Oct 20. PMID 37871604
- [Result] Janjigian YY, Kawazoe A, Bai Y, Xu J, Lonardi S, Metges JP, Yanez P, Wyrwicz LS, Shen L, Ostapenko Y, Bilici M, Chung HC, Shitara K, Qin S, Van Cutsem E, Tabernero J, Luo S, Mahave M, Tang Y, Lowery M, Monteiro MMF, Xu L, Shih CS, Sharan KP, Bhagia P, Rha SY. Pembrolizumab in HER2-Positive Gastric Cancer. N Engl J Med. 2024 Oct 10;391(14):1360-1362. doi: 10.1056/NEJMc2408121. Epub 2024 Sep 14. No abstract available. PMID 39282917
- [Derived] Janjigian YY, Kawazoe A, Yanez P, Li N, Lonardi S, Kolesnik O, Barajas O, Bai Y, Shen L, Tang Y, Wyrwicz LS, Xu J, Shitara K, Qin S, Van Cutsem E, Tabernero J, Li L, Shah S, Bhagia P, Chung HC. The KEYNOTE-811 trial of dual PD-1 and HER2 blockade in HER2-positive gastric cancer. Nature. 2021 Dec;600(7890):727-730. doi: 10.1038/s41586-021-04161-3. Epub 2021 Dec 15. PMID 34912120
- [Derived] Chung HC, Bang YJ, S Fuchs C, Qin SK, Satoh T, Shitara K, Tabernero J, Van Cutsem E, Alsina M, Cao ZA, Lu J, Bhagia P, Shih CS, Janjigian YY. First-line pembrolizumab/placebo plus trastuzumab and chemotherapy in HER2-positive advanced gastric cancer: KEYNOTE-811. Future Oncol. 2021 Feb;17(5):491-501. doi: 10.2217/fon-2020-0737. Epub 2020 Nov 10. PMID 33167735
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26254&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per protocol, response or progression for participants in the Japan-specific SOX (S-1 plus oxaliplatin) Cohort and for participants in the second course of pembrolizumab were not counted towards efficacy analysis, and adverse events for participants during the second course of pembrolizumab were not counted towards safety analysis.
Groups:
- Global Pembrolizumab + Standard of Care First Course: Participants received 200 mg pembrolizumab intravenously (IV) every 3 weeks (Q3W) plus trastuzumab (8 mg/kg loading dose, 6 mg/kg maintenance thereafter) IV Q3W in combination with cisplatin plus 5-fluorouracil (FP) or capecitabine/oxaliplatin (CAPOX) chemotherapy. Eligible participants from the Global Cohort Pembrolizumab + Standard of Care who stopped initial course of pembrolizumab due to complete response (CR) or who had stable disease (SD), PR, or CR after completion of 35 cycles of pembrolizumab but progressed after discontinuation, initiated a second course of pembrolizumab at the investigator's discretion. Participants received 200 mg pembrolizumab IV every 3 weeks (Q3W) for up to 17 additional cycles (approximately 1 year additional treatment).
- Global Standard of Care: Participants received matched placebo to pembrolizumab IV Q3W plus trastuzumab (8mg/kg loading dose, 6mg/kg maintenance thereafter) IV Q3W in combination with FP or CAPOX chemotherapy.
Period: Overall Study
Arm/Group | Global Pembrolizumab + Standard of Care First Course | Global Standard of Care | Japan Pembrolizumab + Trastuzumab + S-1 Plus Oxaliplatin | Japan Trastuzumab + S-1 Plus Oxaliplatin
Started | 350 | 348 | 20 | 20
Treated | 350 | 346 | 20 | 20
Received Second Course of Pembrolizumab | 11 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 350 | 348 | 20 | 20
Not completed — Death | 266 | 286 | 14 | 17
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 3 | 0 | 0
Not completed — Participants Ongoing | 83 | 58 | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Global Pembrolizumab + Standard of Care First Course: Participants received 200 mg pembrolizumab IV every 3 weeks (Q3W) plus trastuzumab (8 mg/kg loading dose, 6 mg/kg maintenance thereafter) IV Q3W in combination with FP or CAPOX chemotherapy. Eligible participants from the Global Cohort Pembrolizumab + Standard of Care who stopped initial course of pembrolizumab due to complete response (CR) or who had stable disease (SD), PR, or CR after completion of 35 cycles of pembrolizumab but progressed after discontinuation, initiated a second course of pembrolizumab at the investigator's discretion. Participants received 200 mg pembrolizumab IV every 3 weeks (Q3W) for up to 17 additional cycles (approximately 1 year additional treatment).
- Total: Total of all reporting groups
Arm/Group | Global Pembrolizumab + Standard of Care First Course | Global Standard of Care | Japan Pembrolizumab + Trastuzumab + S-1 Plus Oxaliplatin | Japan Trastuzumab + S-1 Plus Oxaliplatin | Total
Number analyzed (Participants) | 350 | 348 | 20 | 20 | 738
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.4 (11.8) | 61.7 (10.8) | 66.1 (12.8) | 64.1 (6.8) | 61.2 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 68 | 3 | 5 | 142
  Male | 284 | 280 | 17 | 15 | 596
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38 | 45 | 1 | 1 | 85
  Not Hispanic or Latino | 309 | 293 | 19 | 19 | 640
  Unknown or Not Reported | 3 | 10 | 0 | 0 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 6 | 0 | 0 | 11
  Asian | 119 | 121 | 20 | 20 | 280
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 0 | 0 | 4
  White | 218 | 212 | 0 | 0 | 430
  More than one race | 6 | 5 | 0 | 0 | 11
  Unknown or Not Reported | 0 | 2 | 0 | 0 | 2
Geographic Region [Count of Participants; unit: Participants] — Per protocol, participants in the Global Cohort were stratified by geographic region using the following categories: Western Europe/Israel/North America/Australia; Asia; and Rest of World. Per protocol, participants in the Japan-specific SOX Cohort were not stratified by geographic region.
  Participants
    Western Europe/Israel/North America/Australia | 113 | 111 | 0 | 0 | 224
    Asia | 118 | 119 | 0 | 0 | 237
    Rest of the World | 119 | 118 | 0 | 0 | 237
    Japan | 0 | 0 | 20 | 20 | 40
Programmed Cell Death Ligand 1 (PD-L1) Combined Positive Score (CPS) Status at Baseline [Count of Participants; unit: Participants] — PD-L1 combined positive score (CPS) at baseline was determined by immunohistochemistry (IHC) using an archival tumor sample. The number of participants with CPS<1 and CPS≥1 at baseline is presented. Participants with a CPS<1 were classified as PD-L1 negative and participants with a CPS≥1 were classified as PD-L1 positive. Per protocol, participants in both the Global Cohort and Japan-specific SOX Cohort were stratified by PD-L1 CPS status at baseline.
  Participants
    CPS≥1 | 298 | 296 | 16 | 17 | 627
    CPS<1 | 52 | 52 | 4 | 3 | 111
Chemotherapy Regimen [Count of Participants; unit: Participants] — Per protocol, participants in the Global Cohort were stratified by chemotherapy regimen. Chemotherapy regimen options were FP: cisplatin plus 5-fluorouracil (5-FU) or CAPOX: capecitabine and oxaliplatin. Per protocol, participants in the Japan-specific SOX Cohort were not stratified by chemotherapy regimen.
  Participants
    FP (cisplatin plus 5 fluorouracil) | 53 | 49 | 0 | 0 | 102
    CAPOX (capecitabine and oxaliplatin) | 297 | 299 | 0 | 0 | 596
    SOX (S-1 plus oxaliplatin) | 0 | 0 | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Per RECIST 1.1 Assessed by BICR
Description: PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 as assessed by BICR or death due to any cause, whichever occurs first. Per RECIST 1.1, progressive disease (PD) is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression. PFS was determined for first course pembrolizumab in the Global Cohort. Per statistical analysis plan, participants in the Japan-specific SOX Cohort were not included in the efficacy analysis.
Time Frame: Up to 46 months
Population: All randomized Global Cohort participants in the Pembrolizumab First Course arm and SOC arm were included in this analysis. Per statistical analysis plan, participants in the Japan-specific SOX Cohort were not included in the efficacy analysis.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Global Pembrolizumab + Standard of Care First Course: Participants received 200 mg pembrolizumab IV every 3 weeks (Q3W) plus trastuzumab (8 mg/kg loading dose, 6 mg/kg maintenance thereafter) IV Q3W in combination with FP or CAPOX chemotherapy.
Arm/Group | Global Pembrolizumab + Standard of Care First Course | Global Standard of Care
Number analyzed (Participants) | 350 | 348
Months | 10.0 [8.6 to 12.2] | 8.1 [7.0 to 8.5]
Statistical Analysis 1: Comparison: Global Pembrolizumab + Standard of Care First Course vs Global Standard of Care; PFS in all participants of the Global Pembrolizumab + SOC First Course was compared to PFS in all participants of the Global Standard of Care to address the hypothesis (pembrolizumab in combination with trastuzumab plus chemotherapy is superior to trastuzumab plus chemotherapy alone); Test type: Superiority — The hazard ratio (HR) and its 95% confidence interval (CI) were estimated using a stratified Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by geographic region, PD-L1 status (positive vs. negative) at baseline, and chemotherapy regimen (FP or CAPOX); p = 0.0002, Log Rank; One-sided p-value based on log-rank test stratified by geographic region, PD-L1 status, and chemotherapy regimen with small strata collapsed; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.61 to 0.87] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by geographic region, PD-L1 status, and chemotherapy regimen with small strata collapsed

2. Primary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization to death due to any cause. OS was determined for first course pembrolizumab in the Global Cohort. Per statistical analysis plan, participants in the Japan-specific SOX Cohort were not included in the efficacy analysis.
Time Frame: Up to 63 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Global Standard of Care First Course: Participants received matched placebo to pembrolizumab IV Q3W plus trastuzumab (8mg/kg loading dose, 6mg/kg maintenance thereafter) IV Q3W in combination with FP or CAPOX chemotherapy.
Arm/Group | Global Pembrolizumab + Standard of Care First Course | Global Standard of Care First Course
Number analyzed (Participants) | 350 | 348
Months | 20.0 [17.8 to 22.1] | 16.8 [14.9 to 18.7]
Statistical Analysis 1: Comparison: Global Pembrolizumab + Standard of Care First Course vs Global Standard of Care First Course; OS in all participants of the Global Pembrolizumab + SOC First Course was compared to PFS in all participants of the Global Standard of Care to address the hypothesis (pembrolizumab in combination with trastuzumab plus chemotherapy is superior to trastuzumab plus chemotherapy alone); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0040, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.67 to 0.94] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Objective Response Rate (ORR) Per RECIST 1.1 Assessed by BICR
Description: ORR is defined as the percentage of participants who have a Complete Response ([CR], disappearance of all evidence of disease) or Partial Response ([PR], regression of measurable disease and no new sites) per RECIST 1.1 as assessed by blinded independent central review (BICR). ORR was determined for first course pembrolizumab in the Global Cohort. Per statistical analysis plan, participants in the Japan-specific SOX Cohort were not included in the efficacy analysis.
Time Frame: Up to 63 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Global Pembrolizumab + Standard of Care First Course | Global Standard of Care First Course
Number analyzed (Participants) | 350 | 348
Percentage of Participants | 72.6 [67.6 to 77.2] | 60.1 [54.7 to 65.2]
Statistical Analysis 1: Comparison: Global Pembrolizumab + Standard of Care First Course vs Global Standard of Care First Course; ORR in all participants of the Global Pembrolizumab + SOC First Course was compared to PFS in all participants of the Global Standard of Care to address the hypothesis (pembrolizumab in combination with trastuzumab plus chemotherapy is superior to trastuzumab plus chemotherapy alone); Test type: Superiority — The difference in percentage and its 95% confidence interval (CI) were estimated using the Miettinen & Nurminen method stratified by geographic region, PD-L1 status (positive vs. negative) at baseline, and chemotherapy regimen (FP or CAPOX); p = 0.00020, Stratified Miettinen and Nurminen Method — One-sided p-value for testing. H0: difference in % = 0 versus H1: difference in % > 0; Difference in Percentage = 12.6, 95% CI 2-sided [5.6 to 19.4]

4. Secondary Outcome: Duration of Response (DOR) Per RECIST 1.1 Assessed by BICR
Description: For participants who demonstrate CR or PR, DOR is defined as the time from first response (CR or PR) to subsequent disease progression or death from any cause, whichever occurs first. DOR was determined for first course pembrolizumab in the Global Cohort. Per statistical analysis plan, participants in the Japan-specific SOX Cohort were not included in the efficacy analysis.
Time Frame: Up to 63 months
Population: All randomized Global Cohort participants in the Pembrolizumab First Course arm and SOC arm and who had CR or PR per RECIST 1.1 as assessed by BICR were included in this analysis. Per statistical analysis plan, participants in the Japan-specific SOX Cohort were not included in the efficacy analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Global Pembrolizumab + Standard of Care First Course | Global Standard of Care First Course
Number analyzed (Participants) | 254 | 209
Months | 11.13 [9.8 to 12.7] | 9.5 [7.2 to 11.2]

5. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a participant that is temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment. The number of participants who experienced an AE is reported for each treatment arm. Per statistical analysis plan, data from the second course of pembrolizumab was not included in the safety analysis.
Time Frame: Up to 63 months
Population: All randomized participants in the Global Cohort Pembrolizumab and SOC arms who received at least 1 dose of treatment, and all participants in the Japan-specific SOX Cohort who received at least 1 dose of treatment were included in this analysis. Per statistical analysis plan, data from the second course of pembrolizumab was not included in the safety analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Global Pembrolizumab + Standard of Care First Course | Global Standard of Care First Course | Japan Pembrolizumab + Trastuzumab + S-1 Plus Oxaliplatin | Japan Trastuzumab + S-1 Plus Oxaliplatin
Number analyzed (Participants) | 350 | 346 | 20 | 20
Participants | 348 | 346 | 20 | 20

6. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to AEs
Description: An AE is any untoward medical occurrence in a participant that is temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment. The number of participants who discontinued study treatment due to an AE is reported for each treatment arm. Per statistical analysis plan, data from the second course of pembrolizumab was not included in the safety analysis.
Time Frame: Up to 63 months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Global Pembrolizumab + Standard of Care First Course | Global Standard of Care First Course | Japan Pembrolizumab + Trastuzumab + S-1 Plus Oxaliplatin | Japan Trastuzumab + S-1 Plus Oxaliplatin
Number analyzed (Participants) | 350 | 346 | 20 | 20
Participants | 150 | 136 | 11 | 11

ADVERSE EVENTS:
Time Frame: Up to 63 months
Description: All-Cause Mortality is reported for all randomized participants. Serious Adverse Events and Other Adverse Events are reported for all participants who received treatment. Per protocol, All Cause Mortality and AEs were reported separately for Global Pembrolizumab + SOC and Global Pembrolizumab + SOC Second Course arms.
Groups:
- Global Pembrolizumab + Standard of Care Second Course: Eligible participants from the Global Cohort Pembrolizumab + Standard of Care who stopped initial course of pembrolizumab due to complete response (CR) or who had stable disease (SD), PR, or CR after completion of 35 cycles of pembrolizumab but progressed after discontinuation, initiated a second course of pembrolizumab at the investigator's discretion. Participants received 200 mg pembrolizumab IV every 3 weeks (Q3W) for up to 17 additional cycles (approximately 1 year additional treatment).
Arm/Group | Global Pembrolizumab + Standard of Care First Course | Global Standard of Care | Japan Pembrolizumab + Trastuzumab + S-1 Plus Oxaliplatin | Japan Trastuzumab + S-1 Plus Oxaliplatin | Global Pembrolizumab + Standard of Care Second Course
All-Cause Mortality (participants affected / at risk) | 264/350 | 288/348 | 14/20 | 17/20 | 3/11
Serious Adverse Events (participants affected / at risk) | 163/350 | 159/346 | 10/20 | 9/20 | 0/11
Other Adverse Events (participants affected / at risk) | 345/350 | 338/346 | 20/20 | 20/20 | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Global Pembrolizumab + Standard of Care First Course (N=350) | Global Standard of Care (N=346) | Japan Pembrolizumab + Trastuzumab + S-1 Plus Oxaliplatin (N=20) | Japan Trastuzumab + S-1 Plus Oxaliplatin (N=20) | Global Pembrolizumab + Standard of Care Second Course (N=11)
Anaemia (Blood and lymphatic system disorders) | 5 (6) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Granulocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prinzmetal angina (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypopituitarism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 4 (6) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 17 (19) | 16 (17) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 6 (6) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 3 (3) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Enterocutaneous fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 4 (6) | 6 (10) | 0 (0) | 0 (0) | 0 (0)
Gastric stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 3 (5) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (5) | 0 (0) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal fibrosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal stent stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 (6) | 5 (7) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 7 (9) | 9 (9) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 5 (5) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Sudden death (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Gallbladder obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatorenal syndrome (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 3 (3) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal oesophagitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection in an immunocompromised host (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 19 (20) | 9 (10) | 2 (2) | 1 (1) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Splenic abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 7 (7) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma site discharge (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transcription medication error (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood fibrinogen decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cortisol decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 1 (1) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 2 (2) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2) | 6 (7) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Immune-mediated arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertebral osteophyte (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer fatigue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Central nervous system lesion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebellar haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Horner's syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychogenic seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device failure (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 6 (6) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prerenal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Global Pembrolizumab + Standard of Care First Course (N=350) | Global Standard of Care (N=346) | Japan Pembrolizumab + Trastuzumab + S-1 Plus Oxaliplatin (N=20) | Japan Trastuzumab + S-1 Plus Oxaliplatin (N=20) | Global Pembrolizumab + Standard of Care Second Course (N=11)
Anaemia (Blood and lymphatic system disorders) | 157 (269) | 159 (257) | 5 (6) | 4 (4) | 2 (4)
Leukopenia (Blood and lymphatic system disorders) | 12 (26) | 23 (46) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 59 (133) | 57 (111) | 1 (2) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 43 (67) | 43 (71) | 0 (0) | 0 (0) | 0 (0)
Hypopituitarism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 36 (42) | 16 (22) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 42 (48) | 41 (63) | 2 (3) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 23 (25) | 27 (30) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 62 (80) | 68 (81) | 8 (8) | 5 (5) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 177 (330) | 152 (295) | 12 (30) | 12 (25) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 24 (27) | 17 (17) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 24 (31) | 23 (23) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 5 (5) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 167 (339) | 164 (323) | 9 (12) | 11 (15) | 2 (2)
Pancreatic fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 39 (61) | 30 (39) | 8 (12) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 114 (199) | 92 (163) | 9 (13) | 5 (7) | 1 (1)
Asthenia (General disorders) | 50 (90) | 65 (112) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 78 (113) | 75 (96) | 5 (7) | 3 (3) | 1 (1)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Malaise (General disorders) | 31 (41) | 26 (32) | 5 (7) | 6 (7) | 0 (0)
Mucosal inflammation (General disorders) | 27 (37) | 26 (35) | 0 (0) | 0 (0) | 1 (2)
Oedema peripheral (General disorders) | 31 (37) | 27 (32) | 4 (4) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 53 (80) | 42 (59) | 2 (3) | 6 (8) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 4 (4) | 6 (6) | 0 (0) | 2 (2) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 5 (7) | 3 (5) | 0 (0) | 0 (0) | 3 (4)
Hypersensitivity (Immune system disorders) | 10 (14) | 6 (8) | 2 (3) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 24 (28) | 10 (10) | 1 (1) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 11 (13) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Pneumonia (Infections and infestations) | 21 (23) | 9 (11) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 9 (9) | 11 (14) | 1 (3) | 2 (2) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 36 (44) | 33 (37) | 3 (4) | 2 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 65 (92) | 47 (80) | 1 (1) | 2 (3) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 85 (136) | 63 (108) | 2 (3) | 2 (4) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 18 (20) | 22 (34) | 0 (0) | 1 (2) | 1 (1)
Blood bilirubin increased (Investigations) | 51 (105) | 33 (81) | 0 (0) | 3 (3) | 1 (1)
Blood creatinine increased (Investigations) | 30 (43) | 14 (18) | 1 (2) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 16 (21) | 13 (33) | 1 (1) | 2 (3) | 0 (0)
Neutrophil count decreased (Investigations) | 98 (258) | 85 (297) | 14 (29) | 11 (27) | 1 (2)
Platelet count decreased (Investigations) | 96 (216) | 97 (216) | 7 (9) | 8 (8) | 1 (1)
Weight decreased (Investigations) | 75 (88) | 64 (72) | 4 (4) | 5 (5) | 0 (0)
White blood cell count decreased (Investigations) | 55 (146) | 42 (162) | 3 (8) | 3 (5) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 111 (169) | 110 (147) | 12 (17) | 6 (7) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 23 (39) | 21 (31) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 54 (90) | 57 (93) | 2 (2) | 4 (4) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 21 (26) | 19 (29) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 53 (87) | 39 (62) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 24 (31) | 14 (18) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 23 (27) | 26 (33) | 0 (0) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 14 (18) | 15 (21) | 2 (2) | 2 (3) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 (35) | 16 (17) | 0 (0) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 22 (23) | 22 (25) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 20 (23) | 12 (16) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 17 (18) | 16 (17) | 9 (10) | 4 (4) | 0 (0)
Headache (Nervous system disorders) | 22 (25) | 21 (25) | 1 (1) | 2 (2) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 65 (80) | 65 (88) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 28 (49) | 23 (28) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 85 (119) | 73 (89) | 14 (21) | 14 (17) | 0 (0)
Insomnia (Psychiatric disorders) | 22 (24) | 16 (17) | 1 (1) | 3 (3) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 2 (3) | 2 (2) | 0 (0) | 1 (1)
Urethral haemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 31 (36) | 20 (20) | 1 (1) | 0 (0) | 1 (1)
Dysaesthesia pharynx (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (4) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 (21) | 12 (15) | 0 (0) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14 (23) | 12 (13) | 2 (2) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 19 (24) | 10 (12) | 3 (4) | 4 (4) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 23 (25) | 15 (15) | 2 (2) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 81 (98) | 78 (93) | 4 (5) | 4 (4) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 31 (35) | 20 (20) | 4 (4) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 30 (33) | 15 (18) | 5 (8) | 2 (2) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 7 (7) | 8 (8) | 2 (2) | 1 (1) | 0 (0)
Xeroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 20 (35) | 17 (20) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

DOCUMENTS (2):
  • Study Protocol (2022-09-08): https://cdn.clinicaltrials.gov/large-docs/26/NCT03615326/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-07): https://cdn.clinicaltrials.gov/large-docs/26/NCT03615326/SAP_001.pdf